CLINICAL TRIAL: NCT05815459
Title: Mobile Observation Of Depression
Acronym: MOOD
Status: Completed | Type: Observational
Sponsor: Emteq Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MOOD
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder; Major Depressive Episode; Bipolar Disorder
Keywords: Digital phenotyping; Emotion; OCOSense; Wearables; Multimodal
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Cases: Participants wear OCOsense during mood induction tasks tracking hedonic, self-reflective and autobiographical processes respectively. Participants also wear OCOsense whilst engaging in simple physical activities.
  Interventions: Device: OCOsense
- Control Cases: Participants wear OCOsense during mood induction tasks tracking hedonic, self-reflective and autobiographical processes respectively. Participants also wear OCOsense whilst engaging in simple physical activities.
  Interventions: Device: OCOsense

INTERVENTIONS:
Device: OCOsense — Volunteers wear OCOsense glasses continuously during testing to monitor biobehavioural responses to tasks

SUMMARY:
The primary aim of this project is to test if OCOsense glasses can function as a digital phenotyping tool derived from behavioural and physiological signals related to facial expression and motion recorded using the glasses.

DETAILED DESCRIPTION:
Assessment of participants living with a DSM5 research diagnosis of Bipolar disorder or Major depressive disorder as well as healthy controls who will be recruited and characterised through precision phenotyping involving cross-sectional assessment of biobehavioural and physiological markers of the symptoms of depression. Correlations between objective (i.e., OCOsense glasses captured) and subjective (i.e., self-reported) symptoms of depression will be measured within as well as across diagnoses. The resulting biobehavioral clusters will form the building block of a digital phenotyping tool based upon the wider spectrum of non-verbal behaviours and physiology defined and affected by the phenotype of depression.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Ability to read & understand English. This is because the majority of our questionnaires are validated in the English language only.
* Able to walk, sit, lay and stand unaided

Clinical cases:

● ≥ 15 on the Patient health Questionnaire-9 (PhQ9) (moderate to severe depression)

Exclusion Criteria:

Healthy control participants:

* Self-reported current or past history (suspected or diagnosed) of any psychiatric condition
* <5 on the Generalised Anxiety Disorder-7 questionnaire (GAD-7)
* <5 on the PhQ-9 (no depression)
* Receiving medication for any psychiatric disorder (excluding fibromyalgia)

All participants:

* < 18 years of age or >40 years of age
* Anatomical constraints that affect fit (e.g. facial disfigurement)
* Facial nerve damage which limits the ability to make facial expressions
* Body Mass Index (BMI) >29.9 which we deem may affect physical mobility

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Convenience sampling of young adults.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The demonstration of a significant association between facial expression-derived objective valence and self-reported subjective mood under controlled exposure | 4 hours
  Measures of facial muscular activation in the corrugator supercilli and zygomaticus major muscles. By comparing the ratio of corrugator to zygomatic muscle activation, the OCOsense glasses will produce:
  - Objective valence at a given time (ratio/intensity of corrugator to zygomatic muscle activation at that time).
The demonstration of a significant association between facial expression derived objective mood and self-reported subjective mood under controlled exposure | 4 hours
  Measures of facial muscular activation in the corrugator supercilli and zygomaticus major muscles. By measuring corrugator and zygomatic muscle activation, the OCOsense glasses will produce:
  - Objective mood during negatively valenced exposures, neutrally valenced exposures and positively valenced exposures described in terms of expression intensity and variability for each exposure.
Identifying physical activity engagement. | 2 hours
  The OCOsense glasses contain Inertial Measurement Units (IMU) sensors. By detecting inertial displacement over time OCOsense will detect:
  - Movement: a measure of movement over a period of time - specifically, how much of the time period is spent (i) stationary, (ii) in motion, (iii) fidgeting, (iv) engaging with a variety of activities of daily living

SECONDARY OUTCOMES:
Investigating the relationship between vocal prosody and self-reported subjective mood | 2 hours
  The OCOsense glasses contain a microphone. By detecting vocal parameters over time OCOsense will detect:
  - the nonsemantic lexical features of speech related to pitch and tone whilst participants verbally recall a positive event in their life or engage with a semi-structured diagnostic interview.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nduka, MA, MD, FRCS, Study Director — Emteq CSO
Locations (1):
- Emteq Labs, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Where possible, fully anonymised data will be hosted on a secure data responsibility. Specific details will be updated.